CLINICAL TRIAL: NCT01200966
Title: Ethanol Response in Essential Tremor: Clinical and Neurophysiological Correlates
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100199; 10-N-0199
Record Dates: First submitted 2010-09-11; First posted 2010-09-14 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-01-04

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; Transcranial Magnetic Stimulation (TMS); Ethanol; Alcohol; Alcohol Clamp; ET
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
Background:

- Essential tremor (ET) is a neurological disorder involving uncontrollable shaking, which over time can interfere with mobility and affect routine aspects of daily living. Several medications are used to treat ET, but these medications are often only partially effective and can have side effects. About two-thirds (66%) of people with ET have some relief from drinking alcohol, which suggests that alcohol affects the part of the brain causing the tremor. However, more research is needed to better understand the effects of alcohol or what areas of the brain might be important in the response.

Objectives:

* To study to what extent alcohol is reducing tremor in a group of patients with essential tremor.
* To use transcranial magnetic stimulation to study the effects of alcohol on essential tremor.

Eligibility:

- Individuals who are at least 21 years of age, have been diagnosed with essential tremor and have tremor in both hands, and can tolerate being off all medications for essential tremor for up to 4 weeks.

Design:

* This study has one screening visit (1 to 2 hours), followed by one study visit (3 to 5 hours). Participants might be asked to also take part in one additional study visit (3 to 5 hours). The maximum period between the study visits is 3 months.
* Participants will be screened with a medical history, physical examination, and blood tests. At this visit, participants will receive information about how to safely taper off their current ET medications before the start of the study.
* Participants must be willing to abstain from drinking any alcohol or caffeine (or consuming foods with caffeine such as chocolate) for at least 2 days before the study visits. Participants must also fast overnight (for at least 8 hours) before the study visits.
* At the first study visit, participants will receive a single drink of alcohol (mixed with a noncaffeinated drink) and will complete movement tests to determine whether the alcohol improves the tremor. Alcohol levels will be monitored throughout the visit.
* At the second study visit, participants will have an electrocardiogram to measure heart electrical activity and determine if they are able to safely have transcranial magnetic stimulation. Participants will then receive an intravenous infusion of alcohol and complete questionnaires during the infusion to provide information about its effects. Then, transcranial magnetic stimulation will be used to study brain electrical activity, as well as muscle movements and tremor activity, while under the influence of the alcohol infusion.
* After each study visit, participants will remain at the clinical center until the effects of the alcohol have worn off. Participants will be able to resume taking their ET medications after the end of the study.

DETAILED DESCRIPTION:
OBJECTIVE:

The objective of this study is to investigate the clinical and electrophysiological correlates of the ethanol response in suppressing the tremor amplitude in patients with essential tremor (ET).

STUDY POPULATION:

85 patients with clinically diagnosed ET according to published diagnostic criteria will be entered into study phase 1. From the groups of participants in study phase 1, 12 responders and 12 non-responders will be invited back to participate in study phase 2.

DESIGN:

In study phase 1, the response to ethanol will be measured by a quantitative and qualitative approach using Essential Tremor (ET) spiral analysis during a standardized oral ethanol challenge. The clinical response will be correlated to breath-alcohol levels. Participants of study phase 1 will be selected based on their rate of response - dichotomized into a group of responders vs. non-responders - for study phase 2, during an IV ethanol challenge, brain excitability will be tested using transcranial magnetic stimulation (TMS).

OUTCOME MEASURES:

As the primary outcome parameter of study phase 1, we will determine the patients who respond to ethanol by tremor reduction versus patients without reduction of tremor intensities, as measured using spiral analysis of the dominant hand. Criterion for response will be operationally defined in a dichotomized fashion as reduction of tremor intensities, larger than the known diurnal variation of ET. Therefore, a patient will be considered a responder, if spirographic tremor amplitudes decrease by 35% or more at the time-point 60 minutes after an oral ethanol administration, as compared to baseline. As secondary outcome parameters, spiral data from the non-dominant hand, as well as clinical rating scales and breath alcohol levels will be measured to correlate objective with subjective ratings of ethanol effect in ET.

In study phase two, changes of short intracortical inhibition (SICI), known to be mediated by GABAA, will be analyzed using TMS and compared between responders and non-responders before and during a constant iv administration of ethanol. Secondary outcome parameters include the measurement of changes of GABAB-mediated paradigms such as long intracortical inhibition (LICI), cortical silent period (CSP), intracortical facilitation (ICF), motor evoked potential recruitment curve as well as TMS-measures of cerebellar inhibition.

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosis of essential tremor with bilateral hand tremor as the predominant feature

Unequivocal spirographic tremor of both hands on screening examination

Subjects must be willing and safely able to comply with the study protocol and therefore abstain from any medication for the treatment of tremor for a period of at least 5 plasma half-lives of the individual drug prior to study participation. (For Propranolol/Inderal , Gabapentin/Neurontin this will be 1 day; for Primidone/Mysoline : 26 days).

Subjects must be willing to refrain from alcohol and drinks or food containing caffeine starting 48 hours prior to the study visit(s)

EXCLUSION CRITERIA:

Patients with any other significant pathological finding in the neurological examination other than typical symptoms of ET

Acute or chronic severe medical conditions which would preclude the subject from participating (e.g., severe heart disease NYHA grade 3 or 4, renal failure, hepatic failure, lung disease, uncontrolled hyperthyroidism)

Subjects with active or past alcohol abuse or dependence

Elevated liver function parameters (AST, ALT, GGT), higher than the 1.5 fold upper limit of the normal range (as defined by the NIH Clinical Center Laboratory Medicine Department). The limit for AST therefore will be 51 U/l, for ALT 62 U/L, and GGT 128 U/l.

Female subjects who are pregnant or lactating

Subjects aged < 21 years

Subjects with unable or unwilling to give informed consent

Subjects unable or unwilling to cooperate with study requirements Use of prescription or OTC medications that interact with ethanol or influence brain excitability (e.g. hypnotic, antiepileptic, antipsychotic medication, stimulants, antihistamines, muscle relaxants, etc.).

Known flushing symptoms after alcohol intake or allergy to alcohol.

ADDITIONAL EXCLUSION CRITERIA FOR SUBJECTS ALSO PARTICIPATING IN PHASE 2:

History of seizure disorder or hearing loss

Presence of pacemaker, implanted medical pump, metal plate or metal object in skull or eye.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-08-30; Study Completion 2017-01-04

PRIMARY OUTCOMES:
Phase 1: To objectively determine the rate of ethanol responders vs. non-responders in a prospective sample of ET patients.
Phase 2: To evaluate changes of SICI in responding vs. non-responding ET patients during a continuous ethanol administration

SECONDARY OUTCOMES:
Phase 1: To correlate spirographic and clinical response in both hands with breath-alcohol-levels, acquired using a Breathalyzer at constant intervals after ethanol administration.
Phase 2: To evaluate changes additional TMS measures between groups

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Louis ED, Ottman R, Hauser WA. How common is the most common adult movement disorder? estimates of the prevalence of essential tremor throughout the world. Mov Disord. 1998 Jan;13(1):5-10. doi: 10.1002/mds.870130105. PMID 9452318
- [Background] Deuschl G, Bain P, Brin M. Consensus statement of the Movement Disorder Society on Tremor. Ad Hoc Scientific Committee. Mov Disord. 1998;13 Suppl 3:2-23. doi: 10.1002/mds.870131303. PMID 9827589
- [Background] Wells JN, Shirodkar AV, Knevel AM. Aziridine derivatives as potential monoamine oxidase inhibitors. J Med Chem. 1966 Mar;9(2):195-7. doi: 10.1021/jm00320a009. No abstract available. PMID 5911798